CLINICAL TRIAL: NCT02960750
Title: Effectiveness of a Workplace "Sit Less and Move More" Web-based Program (Walk@WorkSpain) on Occupational Sedentary Behavior, Habitual Physical Activity, Physical Risk Factors for Chronic Disease and Efficiency-related Outcomes in Spanish Office Employees
Brief Title: Effectiveness of a Workplace "Sit Less and Move More" Web-based Program in Spanish Office Employees (Walk@WorkSpain)
Acronym: W@WS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government); University Ramon Llull (Other); University of the Basque Country (UPV/EHU) (Other); University of Vigo (Other); The University of Queensland (Other); University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OR0431+D3009; DEP2009-11472 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación)
Record Dates: First submitted 2016-11-03; First posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Sedentary Lifestyle; Workplace; Quality of Life; Intervention Study
Keywords: workplace; sedentary behavior; physical activity; physical risk factors; mental well-being; presenteeism; work productivity; activity-related energy expenditures
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Had access to the W@WS website program during 19 weeks.
  Interventions: Behavioral: A workplace "sit less and move more" web-based program for Spanish office employees
- Active comparison group (Active Comparator): Maintained habitual behavior.
  Interventions: Behavioral: Active Comparison group

INTERVENTIONS:
Behavioral: A workplace "sit less and move more" web-based program for Spanish office employees — W@WS encourages office employees to progressively 'sit less and move more' during workdays over 19 weeks. During the first 8 weeks (ramping phase), tips are provided every two weeks to break occupational sitting time through incidental movement during work tasks, introduce short walks (5-10 minutes) during morning/afternoon work breaks and/or commuting time, introduce longer walks at lunchtime and achieve at least 10,000 daily steps as well as increase walking intensity. During weeks 9 to 19, W@WS provides automated guidance with periodic emails encouraging behaviors achieved in the previous phase. Ecological support strategies such as logging daily step counts into a personal account and receiving visual feedback on the achievement of goals are also provided
  Other Names: Walk@WorkSpain; W@WS
  Arms: Intervention group
Behavioral: Active Comparison group — The Active Comparison group maintained habitual behavior. The A-CG was given a pedometer and a paper diary to register daily step counts and self-reported sitting time throughout the intervention.
  Other Names: A-CG
  Arms: Active comparison group

SUMMARY:
This study assesses the short and mid-term impacts of a workplace web-based intervention (Walk@WorkSpain, W@WS) on self-reported occupational sitting time, step counts, activity-related energy expenditure, physical risk factors for chronic disease and efficiency-related outcomes in Spanish office employees. Half of participants had access to the W@WS website program while the other half was asked to maintain habitual behaviour.

DETAILED DESCRIPTION:
Rising numbers of people have to sit for long hours every day especially for work and transport (3401184). This sedentary pattern that has been detrimentally associated with obesity and cardiovascular disease markers (4604082). However, replacing as little as 10 minutes of sedentary time with the same amount of light or moderate physical activity is associated with substantial health benefits (i.e. reduction of the metabolic syndrome) (26635358).

Because eighty percent of adults in developed countries spend one third of their working day doing sedentary, desk-based tasks (24603203) -representing a high exposure to this established health risk- displacing occupational sitting with physical activity may be a feasible option for improving office employees´ health and therefore public health (26984326).

In this context, there is a need to develop and evaluate translational research, based on theoretically-derived strategies, that can be successfully embedded into workplaces (26984326).

ELIGIBILITY:
Inclusion Criteria:

* Office employees (university administrative and academic staff) with low and moderate physical activity levels (0 to 3,000 MET·min·wk-1 according to the International Physical Activity Questionnaire)

Exclusion Criteria:

* Highly active office employees (>3,000 MET·min·wk-1 according to the International Physical Activity Questionnaire)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline occupational sitting time (minutes/day) at post-intervention (19 weeks) and two months follow-up. | Baseline,19 weeks, two months follow-up
  A paper diary log assessed self-reported occupational sitting time.
Change from baseline step counts (steps/day) at post-intervention (19 weeks) and two months follow-up | Baseline,19 weeks, two months follow-up
  A pedometer (Yamax 200) assessed daily step counts

SECONDARY OUTCOMES:
Change from baseline waist circumference (cms) at post-intervention (19 weeks) and two months follow-up | Baseline,19 weeks, two months follow-up
  A flexible steel tape (Seca 203) assessed waist circumference
Change from baseline body mass index (kgs/m-2) at post-intervention (19 weeks) and two months follow-up | Baseline, 19 weeks, two months follow-up
  An electronic scale (Seca 899/217) assessed body weight and height to calculate BMI.
Change from baseline blood pressure (mmHg) at post-intervention (19 weeks) and two months follow-up | Baseline, 19 weeks, two months follow-up
  A digital automatic blood pressure monitor (Omron M7) assessed blood pressure.
Change from baseline mental well-being (WEMWBS scale scores) at post-intervention (19 weeks) and two months follow-up | Baseline, 19 weeks, two months follow-up
  The Warwick-Edinburg Mental Well-Being Scale (WEMWBS) assessed mental well-being
Change from baseline presenteeism (WLQ scores) at post-intervention (19 weeks) and two months follow-up | Baseline, 19 weeks, two months follow-up
  The Work Limitations Questionnaire (WLQ) assessed presenteeism.
Change from baseline % work productivity loss (WLQ index score) at post-intervention (19 weeks) and two months follow-up | Baseline, 19 weeks, two months follow-up
  The Work Limitations Questionnaire (WLQ) assessed % of work productivity loss
Change from baseline activity-related energy expenditure (METs-min/week) at post-intervention (19 weeks) and two months follow-up. | Baseline, 19 weeks, two months follow-up
  The International Physical Activity Questionnaire (IPAQ) short form assessed activity-related energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Anna Puig-Ribera, Exercise and Health Sciences, Principal Investigator — University of Vic - Central University of Catalonia
Locations (4):
- Spain (4):
  - University Ramon Llull, Barcelona, Barcelona
  - University of Vic-Central University of Catalonia, Vic, Barcelona
  - University of Vigo, Pontevedra, Galicia
  - Vasque Country University, Vitoria-Gasteiz, Vasque Country

REFERENCES:
- [Result] Mailey EL, Rosenkranz SK, Casey K, Swank A. Comparing the effects of two different break strategies on occupational sedentary behavior in a real world setting: A randomized trial. Prev Med Rep. 2016 Aug 9;4:423-8. doi: 10.1016/j.pmedr.2016.08.010. eCollection 2016 Dec. PMID 27583200
- [Result] De Cocker K, De Bourdeaudhuij I, Cardon G, Vandelanotte C. The Effectiveness of a Web-Based Computer-Tailored Intervention on Workplace Sitting: A Randomized Controlled Trial. J Med Internet Res. 2016 May 31;18(5):e96. doi: 10.2196/jmir.5266. PMID 27245789
- [Result] Eng JY, Moy FM, Bulgiba A. Impact of a Workplace Health Promotion Program on Employees' Blood Pressure in a Public University. PLoS One. 2016 Feb 3;11(2):e0148307. doi: 10.1371/journal.pone.0148307. eCollection 2016. PMID 26840508
- [Result] Shrestha N, Kukkonen-Harjula KT, Verbeek JH, Ijaz S, Hermans V, Bhaumik S. Workplace interventions for reducing sitting at work. Cochrane Database Syst Rev. 2016 Mar 17;3(3):CD010912. doi: 10.1002/14651858.CD010912.pub3. PMID 26984326
- [Result] Cunningham CC, Hager LP. Crystalline pyruvate oxidase from Escherichia coli. II. Activation by phospholipids. J Biol Chem. 1971 Mar 25;246(6):1575-82. No abstract available. PMID 4323230
- [Result] Dube B, Agarwal SP, Gupta MM, Chawla SC. Congenital deficiency of fibrinogen in two sisters. A clinical and haematological study. Acta Haematol. 1970;43(2):120-7. doi: 10.1159/000208721. No abstract available. PMID 4986191
- [Result] Shrager RI, Cohen JS, Heller SR, Sachs DH, Schechter AN. Mathematical models for interacting groups in nuclear magnetic resonance titration curves. Biochemistry. 1972 Feb 15;11(4):541-7. doi: 10.1021/bi00754a010. No abstract available. PMID 5011963
- [Result] Lofgren PA, Warner RG. Relationship of dietary caloric density and certain blood metabolites to voluntary feed intake in mature wethers. J Anim Sci. 1972 Dec;35(6):1239-47. doi: 10.2527/jas1972.3561239x. No abstract available. PMID 4647454
- [Derived] Puig-Ribera A, Bort-Roig J, Gine-Garriga M, Gonzalez-Suarez AM, Martinez-Lemos I, Fortuno J, Martori JC, Munoz-Ortiz L, Mila R, Gilson ND, McKenna J. Impact of a workplace 'sit less, move more' program on efficiency-related outcomes of office employees. BMC Public Health. 2017 May 16;17(1):455. doi: 10.1186/s12889-017-4367-8. PMID 28511642
- Available data/document: Clinical Study Report: 4382156 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4382156/?report=classic
- Available data/document: Clinical Study Report: 4323230 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4323230/?report=classic
- Available data/document: Clinical Study Report: 4266209 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4266209/